CLINICAL TRIAL: NCT01476254
Title: Respiratory Complications After Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Anne Kathrine Staehr, Research Assistant, Herlev Hospital
Other Study IDs: RESP-1
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Pulmonary Atelectasis; Respiratory Insufficiency; Pneumonia
Keywords: Postoperative pulmonary complications; Laparoscopic surgery
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Insufficiency; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cholecystectomy: Women scheduled for laparoscopic cholecystectomy
- Hysterectomy: Women scheduled for laparoscopic hysterectomy

SUMMARY:
The purpose of this study is to describe the magnitude of respiratory complications after laparoscopic hysterectomy and cholecystectomy.

DETAILED DESCRIPTION:
The purpose of this study is to describe change in pulmonary function and incidence of respiratory complications after laparoscopic surgery.

The investigators will include 60 women scheduled for laparoscopic hysterectomy or cholecystectomy. The investigators will measure the pulmonary function by different methods during and for 2 hours after surgery. Moreover, the incidence of respiratory complications including pneumonia, respiratory failure and radiologically verified atelectasis will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Women
* > 45 years old
* Scheduled for laparoscopic cholecystectomy or laparoscopic hysterectomy

Exclusion Criteria:

* Weight < 50 kg
* Pregnant or nursing
* Cardiac failure
* Renal failure
* Inability to breath through a facial mask
* Inability to give informed consent
* Inability to keep arterial oxygen saturation above 90% without supplemental oxygen

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective laparoscopic surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Arterial oxygen tension 2 hours after surgery | 2 hours after end of surgery
  Change in arterial oxygen tension 2 hours after surgery

SECONDARY OUTCOMES:
Oxygenation index 2 hours after surgery | 2 hours after end of surgery
  Change in oxygenation index (PaO2/FiO2) 2 hours after surgery
FEV1 and FVC 2 hours after surgery | 2 hours after end of surgery
  Change in FEV1 and FVC 2 hours after surgery
Pulmonary shunt 2 hours after surgery | 2 hours after end of surgery
  Change in pulmonary shunt 2 hours after surgery
Ventilation-perfusion ratio 2 hours after surgery | 2 hours after end of surgery
  Change in ventilation-perfusion ratio from baseline to 2 hours after surgery
Arterial oxygen saturation 2 hours after surgery | 2 hours after surgery
  Change in arterial oxygen saturation 2 hours after surgery
Respiratory frequency 2 hours after surgery | 2 hours after surgery
  Change in respiratory frequency 2 hours after surgery
Oxygen supplement at discharge from the postanesthesia care unit | At discharge from the postanesthesia care unit, which will be approximately 2 hours after surgery
  The proportion of patients who received oxygen supplement at discharge from the postanesthesia care unit in order keep arterial oxygen saturation above 93%
Connection between pulmonary shunt and need for oxygen supplement | 2 hours postoperatively and at discharge from the postanesthesia care unit
  The connection between pulmonary shunt 2 hours after surgery and need for oxygen supplement at discharge from the postanesthesia department in order to keep peripheral oxygen saturation above 93%.
FEV1 and FVC 24 hours after surgery | 24 hours after surgery
  Change in FEV1 and FVC 24 hours after surgery
Pulmonary shunt 24 hours after surgery | 24 hours after surgery
  Change in pulmonary shunt 24 hours after surgery
Ventilation-perfusion ratio 24 hours after surgery | 24 hours after surgery
  Change in ventilation-perfusion ratio 24 hours after surgery
Arterial oxygen saturation 24 hours after surgery | 24 hours after surgery
  Change in arterial oxygen saturation 24 hours after surgery
Respiratory frequency 24 hours after surgery | 24 hours after surgery
  Change in respiratory frequency 24 hours after surgery
Length of stay | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Length of stay at the hospital
Pneumonia | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Incidence of pneumonia from surgery to discharge from hospital
Respiratory failure after surgery | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Incidence of respiratory failure from surgery to discharge from hospital
Atelectasis | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Incidence of radiologically verified atelectasis from surgery to discharge from hospital
High temperature | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Incidence of a high temperature ( above 38 degrees celsius) from surgery to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mona R Gätke, M.D. Ph.D., Study Chair — Department of Anesthesia, Herlev Hospital, University of Copenhagen; Anne K Staehr, M.D., Principal Investigator — Department of Anesthesia, Herlev Hospital, University of Copenhagen
Locations (2):
- Denmark (2):
  - Department of Anesthesia, Herlev Hospital, Herlev
  - Department of Anesthesia, Hillerød Hospital, Hillerød